CLINICAL TRIAL: NCT04451395
Title: Investigating Pathways Between Maternal Nutritional Status, Breastmilk Composition, and Infant Linear Growth in Rural Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Founding Chair, Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-3676-10314
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Breast Milk Collection; Infant Development
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple micronutrients (UNIMMAP composition) (Experimental): The intervention is an oral tablet containing 15 different vitamins and minerals at the UNIMMAP composition (includes 30 mg iron, 400 μg folic acid, 15 mg zinc, 2 mg copper, 65 μg selenium, 800 μg RE vitamin A, 1.4 mg vitamin B1, 1.4 mg vitamin B2, 18 mg niacin, 1.9 mg vitamin B6, 2.6 μg vitamin B12, 70 mg vitamin C, 5 μg vitamin D, 10 mg vitamin E and 150 μg iodine). Each tablet is small (approximately 10 mm diameter) and has been procured using the UNICEF supply catalogue. A single MMN supplementation dose will consist of a single tablet..The supplement is provided within the parent trial.
  Other Name: UNICEF, Micronutrient tabs, pregnancy/PAC-1000
  Interventions: Dietary Supplement: Multiple micronutrients (UNIMMAP composition)
- Standard of care (No Intervention): Daily iron and folic acid supplementation provided through the existing public health system.

INTERVENTIONS:
Dietary Supplement: Multiple micronutrients (UNIMMAP composition) — The intervention is an oral tablet containing 15 different vitamins and minerals at the UNIMMAP composition (includes 30 mg iron, 400 μg folic acid, 15 mg zinc, 2 mg copper, 65 μg selenium, 800 μg RE vitamin A, 1.4 mg vitamin B1, 1.4 mg vitamin B2, 18 mg niacin, 1.9 mg vitamin B6, 2.6 μg vitamin B12, 70 mg vitamin C, 5 μg vitamin D, 10 mg vitamin E and 150 μg iodine). Each tablet is small (approximately 10 mm diameter) and has been procured using the UNICEF supply catalogue. A single MMN supplementation dose will consist of a single tablet.
  Other Name: UNICEF, Micronutrient tabs, pregnancy/PAC-1000
  Arms: Multiple micronutrients (UNIMMAP composition)

SUMMARY:
Breastmilk is considered optimal for infant growth and development. However, evidence suggests that breastmilk composition can vary according to maternal nutritional status. Among women in Pakistan, there is a high burden of undernutrition and micronutrient deficiencies. As well, the prevalence of early stunting among Pakistani infants is high. Using a hypothesized pathway model, this study will assess pathways between maternal nutritional status, breastmilk composition, and infant linear growth. This is a substudy to the Matiari emPowerment and Preconception Supplementation (MaPPS) Trial (ClinicalTrials.gov Identifier: NCT03287882).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the MaPPS Trial
* Mothers must report practicing exclusive or predominant breastfeeding (i.e., breastmilk only or breastmilk and non-nutritive feeds only)
* The infant must be term-born (>37 weeks gestation)
* Infant must be 3 months ± 30 days old at the time of recruitment
* Mothers must be willing to provide a complete breastmilk expression from one breast
* Intervention arm only: mother reports compliance with study-administered MMN supplements at least 50% of the time (i.e., 4 out of 7 days per week)
* Able to provide informed consent

Exclusion Criteria:

* Mother reports mixed feeding in her infant with nutritive feeds (i.e., any provision of formula or animal milk)
* The infant was born preterm (earlier than 37 weeks gestation)
* Mother does not wish to provide a complete breast expression of one breast
* Intervention arm: mother reports compliance with MMN supplements <50% of the time

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 196 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal BMI | 3 months postpartum
Maternal dietary diversity score | 3 months postpartum
  Minimum score: 0, maximum score: 10
Maternal hemoglobin concentration | 3 months postpartum
Maternal supplement adherence | 3 months postpartum
  Determined by report (options: 0, 25, 50, 75, or 100%)
Breastmilk macronutrient composition | 3 months postpartum
Breastmilk micronutrient composition | 3 months postpartum
Infant length | 3 months postpartum

SECONDARY OUTCOMES:
Infant weight | 3 months postpartum
Infant middle-upper arm circumference | 3 months postpartum
Infant head circumference | 3 months postpartum
Breastmilk bioactive composition | 3 months postpartum
Breastmilk microbiome | 3 months postpartum
Infant microbiome | 3 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Matiari Research and Training Centre, Matiari, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Please contact the Primary Investigator directly for more details.

REFERENCES:
- [Derived] Baxter JB, Wasan Y, Daniel AI, Begum K, Hussain A, Iqbal J, Aufreiter S, Beggs MR, Duan L, Greco A, Huang C, Soofi S, Bandsma RH, Bhutta ZA, O'Connor DL. Maternal multiple micronutrient supplementation in rural Pakistan increased some milk micronutrient concentrations, but not infant growth, at three-months postpartum: a randomized controlled trial substudy. Am J Clin Nutr. 2025 Jul;122(1):174-184. doi: 10.1016/j.ajcnut.2025.05.019. Epub 2025 May 21. PMID 40409469